CLINICAL TRIAL: NCT03824743
Title: Impact of Balanced Crystalloids in Obstetric Hemorrhage: A Prospective Cohort Study
Brief Title: Balanced Crystalloids in Postpartum Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Leopoldo Ferrer, Principal investigator, Fundación Santa Fe de Bogota
Other Study IDs: CCEI-9813-2018
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Ringer's Lactate; Plasma-lyte 148

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lactate Ringer: Patients managed with Ringer Lactate
  Interventions: Drug: Lactate Ringer
- Plasma-Lyte: Patients managed with Plasma-Lyte
  Interventions: Drug: Plasma-lyte

INTERVENTIONS:
Drug: Lactate Ringer — Patients managed with Lactate Ringer and obstetric hemorrhage
  Other Names: Cristalloids
  Groups: Lactate Ringer
Drug: Plasma-lyte — Patients managed with Plasma-Lyte and obstetric hemorrhage
  Other Names: Balanced cristalloids
  Groups: Plasma-Lyte

SUMMARY:
Introduction:

Obstetric hemorrhage is the most feared complication that can occur during childbirth and continues to be the leading cause of death in pregnant women worldwide, about 7 women die every hour in the world. This is defined as an accumulated loss of blood of more than 1000 mL with signs and symptoms of hypovolemia within 24 hours of the birth process. The main objective of resuscitation in these patients is precisely to reduce the deleterious effects that are generated from the depletion of volume and the altered capacity of oxygen transport. The current debate focuses on the safety and efficacy of each particular liquid during resuscitation and on improving long-term patient outcomes. At present, there is no conclusive evidence on the impact at the level of acid-base status, hydroelectrolytic balance and potential kidney injury with respect to the use of balanced solutions such as Plasma-Lyte or Ringer's Lactate.

Objective:

To determine the differences in the volume of liquids and blood products required with the use of balanced crystalloids (Ringer's Lactate or Plasma-Lyte) in patients with obstetric hemorrhage in the Hospital Universitario Fundación Santa Fe de Bogotá during 2018 - 2019.

Design, Materials, and methods:

Historical cohort analytical study. All patients over 18 years of age who present an obstetric hemorrhage defined as bleeding> 1000 mL or less associated with signs or symptoms of hemodynamic instability will be included. The most important exclusion criterion is the presence of active infection at the time of the event. Patients will be divided into two groups, those who underwent hydroelectrolytic resuscitation with Plasma-Lyte and Ringer Lactate.

Results and conclusions With this study, we intend to describe the differences in the base acid status measured by arterial gases in patients with obstetric hemorrhage. The aim is to find a relationship between the different groups with clinical outcomes, such as days of ICU stay and hospitalization, blood transfusion requirement, electrolyte disorders, acute kidney injury and survival.

DETAILED DESCRIPTION:
Problem Statement Maternal mortality is a tragic event with great social, economic and legal impact. The incidence rate varies depending on the source, however, it covers 400 cases per 100,000 live births per year. The first cause of death in these patients is obstetric hemorrhage, which generates 150,000 deaths per year in the world. Not being outside of this situation, Bogotá presents a high number of women who present this complication, being the cause of death in 29% of cases in the years 2012 and 2013. Once this problem is identified, multiple strategies have sought to reduce maternal morbidity and mortality, one of the most influential being the "Millennium Development Goals", now called "Sustainable Development Goals". Associated with these, national and regional public policies are developed that seek to raise awareness about the importance of timely and early diagnosis, multidisciplinary and synchronous management among several health areas with the aim of preventing and treating obstetric hemorrhage to avoid fatal outcomes.

Within the prevention and management of obstetric bleeding, there are behaviors that have shown significant impact on outcomes, such as, for example, the administration of uterotonics in the active management of delivery, which reduce the risk of postpartum hemorrhage by up to 50% or the early administration of tranexamic acid, reducing mortality by 30%. However, despite these advances, a fundamental part of the initial handling of support is the volumetric resuscitation with crystalloids and in this field, although there is an indication to initiate replenishment of losses it is not clear what type of liquid to use and if any given their characteristics intrinsic can be superior to the other.

Justification In clinical practice, the goal of resuscitation is to return to cellular homeostasis. Normal saline has been used for volumetric resuscitation for more than 50 years. However, questions about its suitability have been raised given the association with negative outcomes given its composition and question whether modifications in these would bring better results. Multiple studies associated resuscitation with an unbalanced solution (normal saline) with hyperchloremic acidosis, acute kidney injury and morbidity in general, especially in the critically ill patient.

However, until now the evidence is not conclusive about whether this impact on the base acid state, hydroelectrolytic imbalance, and potential kidney injury is less with "balanced" solutions and generate better clinical results in all scenarios, surgical patients, patients and particularly in hypovolemic shock due to obstetric hemorrhage.

Research question Are there differences in the volume of fluids and blood products to be used in the outcomes of patients with obstetric hemorrhage with the use of balanced crystalloids (Lactate Ringer or Plasma-Lyte) at the Hospital Universitario Santa Fe de Bogotá during the years 2018 - 2019?

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of obstetric hemorrhage (> 1000 mL). Over 18 years.

Exclusion Criteria:

* Patients with incomplete clinical history.
* Patients with active infections.
* Patients with a history of blood dyscrasias.
* Patients with known kidney disease.
* Patient with previous alteration of the acid-base status.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Universe population: Patients with obstetric hemorrhage in the Hospital Universitario Fundación Santa Fe de Bogotá.
  Study population: Patients with obstetric hemorrhage at the Hospital Universitario Fundación Santa Fe de Bogotá that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Differences in the use of fluids and blood products | 2018 - 2019
  Differences in the use of fluids and blood products with the use of balanced crystalloids in obstetric hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo E Ferrer, M.D., Principal Investigator — Hospital Universitario Fundación Santa Fe de Bogotá
Locations (1):
- Hospital Universitario Fundación Santa Fe de Bogotá, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided